CLINICAL TRIAL: NCT07381361
Title: A Randomized Controlled Trial Comparing the Efficacy of Photobiomodulation Therapy and Alpha-Lipoic Acid in the Treatment of Burning Mouth Syndrome
Brief Title: Photobiomodulation Therapy vs. Alpha-Lipoic Acid in Burning Mouth Syndrome Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lu Jiang (Other)
Responsible Party: Sponsor-Investigator, Lu Jiang, Clinical Professor, Sichuan University
Organization: Sichuan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCHSIRB-D-2025-189-R1
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Burning Mouth Syndrome; Low Level Laser Therapy
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Low-Level Light Therapy; Thioctic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PBMT group (Experimental): Burning mouth syndrome (BMS) patients in PBMT group were provided with BMS disease explanation and psychological counseling. They will receive low-energy laser therapy with an energy density of 5 J/cm² and a power of 0.1/0.5 W for a consecutive period of 2 weeks, 5 days per week.
  Interventions: Other: Low Level Laser Therapy
- ALA group (Active Comparator): Burning mouth syndrome (BMS) patients in the ALA group were provided with BMS disease explanation and psychological counseling. Then they took α-lipoic acid (ALA) 3 times a day, after meals, 200 mg each time, for 2 consecutive weeks.
  Interventions: Drug: Alpha Lipoic Acid

INTERVENTIONS:
Other: Low Level Laser Therapy — Energy density: 5 J/cm² Power: 0.1/0.5 W Course of treatment: 2 consecutive weeks, 5 days per week.
  Other Names: PBMT; LLLT; Photobiomodulation Therapy
  Arms: PBMT group
Drug: Alpha Lipoic Acid — Dosage: 600-800 mg ALA Course of treatment: 2 consecutive weeks, 3 times per day
  Arms: ALA group

SUMMARY:
The aim of this study was to evaluate the efficacy of photobiomodulation therapy and alpha-lipoic acid in the treatment of burning mouth syndrome by symptom assessment with visual analogue scale.

DETAILED DESCRIPTION:
Burning mouth syndrome (BMS), hereinafter referred to as BMS, also known as glossodynia, oral mucosal dysesthesia, and other terms, is a type of neurosis. Its prevalence is approximately 0.7%-8%. Currently, the etiology and pathophysiology of BMS are not yet clear, and there is no known cure. Clinical treatment aims to alleviate patients' subjective symptoms, employing drug therapies (such as rinsing with 2%-4% sodium bicarbonate solution, oryzanol, methylcobalamin, alpha-lipoic acid, etc.), or combining cognitive behavioral therapy and removal of local irritants (such as dental calculus), but the therapeutic effects are limited.

Photobiomodulation therapy (PBMT), also known as low-level laser therapy (LLLT), is a therapeutic method that induces a series of physiological effects in cells, tissues, animals, and humans through the irradiation of specific wavelengths of red or near-infrared light. Research indicates that PBMT can alleviate the pain intensity in patients with BMS through its photobiological effects. Research has shown that photobiomodulation therapy can alleviate the pain of patients with burning mouth syndrome through photobiological effects. Therefore, this research project primarily investigates the efficacy of PBMT for BMS and the differences in therapeutic effects under different parameter settings by establishing a controlled trial with a low-energy laser treatment group and an alpha-lipoic acid control group. Based on the results of the clinical trial, this therapy is intended to be promoted.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years
* Diagnosis of Burning Mouth Syndrome (BMS) according to the 3rd edition of the International Classification of Headache Disorders (ICHD-3)
* Daily intraoral burning or dysesthesia lasting for more than 2 hours for over 3 months
* Normal oral mucosa and sensory testing
* Condition not better accounted for by another ICHD-3 diagnosis

Exclusion Criteria:

* Other oral mucosal diseases, such as oral leukoplakia or oral lichen planus
* Diabetes with poor blood glucose control
* Hematological diseases
* Pregnancy or lactation
* Severe mental disorders preventing cooperation with treatment
* Heart failure (New York Heart Association class III-IV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline and 2 weeks after intervention or observation
  The Visual Analogue Scale (VAS) will be used to assess the intensity of the patient's pain. The scale ranges from 0 to 10, where 0 represents "no pain" (the best possible outcome) and 10 represents "the worst pain imaginable" (the worst possible outcome). Therefore, higher scores indicate a worse outcome (greater pain intensity). During the interview or telephone follow-up, the patient will be asked to report the number that best describes their pain.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Jiang, MD, Principal Investigator — Sichuan University
Locations (1):
- West China Hospital of Stomatology, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No